CLINICAL TRIAL: NCT04035889
Title: A Randomized, Crossover Pilot Trial of Melatonin for Sleep Disturbance in Adults With Multiple Sclerosis (MS)
Brief Title: Melatonin for Sleep in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Riley Bove, MD, Assistant Professor of Neurology, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-27108
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
Keywords: Sleep; Melatonin; Sleep disturbance
MeSH Terms: conditions — Multiple Sclerosis; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants assigned to Group 1 will take 2 weeks of melatonin followed by 2 weeks of placebo
  Interventions: Dietary Supplement: Melatonin; Dietary Supplement: Placebo
- Group 2 (Experimental): Participants assigned to Group 2 will take 2 weeks of placebo followed by 2 weeks of melatonin.
  Interventions: Dietary Supplement: Melatonin; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Participants will start with 0.5 mg tablets of melatonin with the option of switching to an 'escalation dose' of 3 mg if no relief after 3 days.
Dietary Supplement: Placebo — Placebo

SUMMARY:
Many people with MS report sleep disturbances. However, objective data on sleep quality in MS, such as those obtained using actigraphy, remain scant, as do data about optimal therapeutic management. Melatonin is frequently used to improve sleep parameters, both in healthy and neurological populations. Altered melatonin regulation and signaling has been implicated in MS, through observations including (1) MS risk associated with shift work, (2) contribution of melatonin to seasonal risk of MS relapses, and (3) possible reduction of endogenous melatonin levels from exogenous corticosteroid administration.

To the best of our knowledge, no studies have evaluated melatonin vs. placebo as a low-cost, low-risk agent to treat sleep disturbance in MS. To test this, we are conducting a randomized controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-70 with a diagnosis of MS by 2010 McDonald Criteria or CIS (clinically isolated syndrome), who report sleep disturbance as measured by a score >=5 on the Pittsburgh Sleep Quality Index, or more specific insomnia symptoms (a score of >14 on the Insomnia Severity Index) over the past month.
* Participants must be able to read and write English

Exclusion Criteria:

* Individuals with nocturnal asthma, use of melatonin or another sleep agent in the past 2 weeks, women attempting conception, relapse or steroids or infusible disease modifying therapies (DMTs) in prior month.
* Non-English speaking individuals
* Individuals with hypertension, impaired liver function, or seizure disorder
* Individuals with untreated depression, as determined by a score greater than or equal to 8 points on the HADS (Hospital Anxiety and Depression Scale)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Sleep time | 4 weeks
  Total sleep time (time in bed spent sleeping after "lights off")
Sleep quality | 4 weeks
  Sleep quality and sleep disturbances assessed by the Pittsburgh Sleep Quality Index and Insomnia Severity Index

SECONDARY OUTCOMES:
Sleep efficiency | 4 weeks
  Sleep efficiency: % time asleep while in bed after "lights off", averaged for mean nightly sleep efficiency
  Sleep onset latency time: time from "lights off" to sleep

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No